CLINICAL TRIAL: NCT00002714
Title: A PHASE II TRIAL OF EIGHT-WEEK STANFORD V CHEMOTHERAPY PLUS MODIFIED INVOLVED FIELD RADIOTHERAPY IN FAVORABLE, LIMITED STAGE HODGKIN'S DISEASE
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Early-Stage Hodgkin's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: SUMC-G4; CDR0000064550 (Registry Identifier: PDQ (Physician Data Query)); NCI-H96-0805
Record Dates: First submitted 1999-11-01; First posted 2004-04-06 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2001-09

CONDITIONS: Lymphoma
Keywords: stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Bleomycin; Doxorubicin; Etoposide; Mechlorethamine; Prednisone; Vinblastine; Vincristine; Radiotherapy

INTERVENTIONS:
Biological: bleomycin sulfate
Drug: Stanford V regimen
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: mechlorethamine hydrochloride
Drug: prednisone
Drug: vinblastine sulfate
Drug: vincristine sulfate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus radiation therapy in treating patients who have early stage Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the progression-free and overall survival at 5 and 10 years after a short-term Stanford V regimen comprising mechlorethamine, doxorubicin, vinblastine, prednisone, vincristine, bleomycin, and etoposide followed by modified involved-field radiotherapy in patients with favorable, early-stage Hodgkin's disease. II. Determine whether the early and late toxic effects of treatment can be minimized by avoiding staging laparotomy, limiting cumulative doses of chemotherapeutic drugs, and reducing the dose and volume of radiotherapy in these patients. III. Determine the freedom from second disease progression at 5 and 10 years after treatment and treatment-related toxicity in these patients. IV. Determine the quality of life of patients treated with this regimen.

OUTLINE: Patients receive the Stanford V regimen comprising mechlorethamine IV on days 1 and 29; doxorubicin IV and vinblastine IV on days 1, 15, 29, and 43; oral prednisone every other day on days 1-36 followed by tapered doses; vincristine IV and bleomycin IV on days 8, 22, 36, and 50; and etoposide IV on days 15, 16, 43, and 44. Beginning 2 weeks after completion of chemotherapy and when blood counts recover, patients undergo modified involved-field radiotherapy 5 days a week for 3-4 weeks. Quality of life is assessed. Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage I-IIA Hodgkin's disease No lymphocyte predominant disease No stage IA high neck presentation (above the top of the larynx) No mediastinal mass equal to or greater than one-third the maximum intrathoracic diameter on chest x-ray No constitutional (B) symptoms at diagnosis No more than 1 extranodal site of disease

PATIENT CHARACTERISTICS: Age: 16 to 60 Performance status: Not specified Hematopoietic: Granulocyte count at least 2,000/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 2.5 mg/dL Renal: Creatinine no greater than 2 mg/dL Other: No other medical condition that would preclude study therapy HIV negative No other prior malignancy except basal cell skin cancer Not pregnant

PRIOR CONCURRENT THERAPY: No prior therapy for Hodgkin's disease No other concurrent antineoplastic therapy No other concurrent investigational drugs

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 1995-04; Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J. Horning, MD, Study Chair — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States